CLINICAL TRIAL: NCT00396474
Title: Long-Term Metabolic Risk In Small for Gestational Age (SGA) Patients After Growth Hormone Treatment Compared To Matched, Untreated Controls
Brief Title: Safety Study In Patients Who Were Born Small And Short And Were Treated With Growth Hormone To Achieve Normal Height
Status: Withdrawn | Type: Observational
Why Stopped: Study design no longer relevant and no patients were recruited.
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Other Study IDs: A6281279
Record Dates: First submitted 2006-11-06; First posted 2006-11-07 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Infant, Small for Gestational Age
Keywords: Small for gestational age, Insulin Sensitivity Index, growth hormone treatment

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood, serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- SGA patients: Infants born small for SGA who either received GH, no GH, or growth within normal ranges.
  Interventions: Other: post GH treatment observational study

INTERVENTIONS:
Other: post GH treatment observational study — Intravenous glucose tolerance test (IVGTT)

SUMMARY:
The purpose of this study is to demonstrate that insulin sensitivity is not different between growth hormone - treated subjects who are small for gestational age (SGA) and an SGA cohort of subjects matched by gender and body mass index (BMI) who are not treated with growth hormone (GH) and who remain short at final height.

DETAILED DESCRIPTION:
case-control

ELIGIBILITY:
Inclusion Criteria:

* Patients with SGA treated with growth hormone in one of the following Genotropin studies (89-041, 89-070/071, 90-079, 90-080/98-8122-011) for at least 3 years and after having stopped GH treatment for 5-10 years
* Untreated SGA (based on birth weight and/or length below -2 standard deviations [SDs] for gestational age) matched to treated SGA by body mass index (+ or = 10%) and gender:

  * Subjects born SGA with normal final height (within +/- 1.3 SD of their target height); or
  * Subjects born SGA with short stature (height SDs > 1.3 below target at final height).

Exclusion Criteria:

* Known diabetes type 1 or 2, or 1st degree relative of a patient with diabetes type 2
* Familial dyslipidemia

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: SGA Subjects treated or untreated with growth hormone
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-01; Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
To demonstrate, that the Insulin Sensitivity Index is not different between GH treated SGA and SGA cohort matched by gender and BMI and not treated with GH that remained short at final height | 90 days

SECONDARY OUTCOMES:
To demonstrate that blood pressure and lipid profile are not different between GH treated SGA subjects and an SGA cohort matched by gender and BMI and not treated with GH | 90 days
To demonstrate that the ISI is not different between GH treated SGA subjects and an SGA cohort matched by gender and BMI and not treated with GH that achieved normal final height | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer